CLINICAL TRIAL: NCT00476229
Title: Total Lymphoid Irradiation, Thymoglobulin, and Rituximab for Allogeneic Transplantation in Lymphoid Malignancies
Brief Title: Thymoglobulin and Total Lymphoid Irradiation for Hematologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0892
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Lymphoma; Leukemia
Keywords: Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Hodgkin's Lymphoma; Lymphoma; Leukemia; Mycophenolate Mofetil; Tacrolimus; Thymoglobulin; Total Lymphoid Irradiation
MeSH Terms: conditions — Lymphoma; Leukemia; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease | interventions — thymoglobulin; Antilymphocyte Serum; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation + Chemotherapy + BSCT (Experimental): Total Lymphoid Irradiation (2 times) at 80 cGy daily for five days + Thymoglobulin 1.5 mg/kg intravenous 5 days + Rituximab 375 mg/m^2 intravenous on 4 different days + Blood stem cell transplant (BSCT)
  Interventions: Drug: Thymoglobulin; Radiation: Total Lymphoid Irradiation; Procedure: Peripheral Blood Stem Cell Infusion; Drug: Rituximab

INTERVENTIONS:
Drug: Thymoglobulin — 1.5 mg/kg by vein on Days -11 to -7.
  Other Names: Antithymocyte Globulin; ATG
Radiation: Total Lymphoid Irradiation — 80 cGy daily on days -11 to -7 and -4 to 0.
  Other Names: TLI
Procedure: Peripheral Blood Stem Cell Infusion — PBSC infusion administered on day 0.
  Other Names: Blood Stem Cell Transplant; BSCT
Drug: Rituximab — 375 mg/m^2 by vein on days -13, -6, 1, & 8. Only those patients whose tumors express CD20 will receive Rituximab.
  Other Names: Rituxan

SUMMARY:
Primary Objective:

1. To determine whether the primary endpoint: the composite success rate, defined as the proportion of patients who are alive at day 100; and are without grade 3-4 Graft versus Host Disease (GVHD); and are without grade 4 toxicity (unrelated to infection); and have engrafted, is likely to be at least 40%.

Secondary Objectives:

1. To determine the cumulative incidence of chronic graft versus host disease.
2. To determine the overall and disease free survival.

DETAILED DESCRIPTION:
The combination of drugs used for this study will help to weaken your immune system, which may help to allow the donor's blood stem cells to engraft (grow) in your body.

Anti-thymocyte globulin (also called ATG or thymoglobulin) is designed to help reduce the risk of transplant rejection and to help prevent graft versus host disease.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

If you are found to be eligible to take part in this study, you will be admitted to the hospital 12 days before the blood stem cell transplant (BSCT), in order to start the pre-transplant treatments and testing. You will have blood (about 1 tablespoon) drawn for routine tests every day while you are in the hospital (before and after the transplant). After the transplant, this blood will be used to check the status of the transplant and watch for any side effects.

You will receive radiation therapy (total lymphoid irradiation) for a total of 10 days before the planned transplant. Radiation therapy will not be given on the weekends. The last radiation treatment will be on the morning of the day you receive your stem cell transplant.

For a total of 5 days after admission to the hospital, you will also receive ATG. ATG will be given through a catheter (plastic tube) that is placed into the large chest vein. The catheter (called a central venous catheter) will stay in place throughout treatment.

You will receive certain drugs as premedication to try to prevent an allergic reaction to the ATG. These may include drugs like acetaminophen (Tylenol), diphenhydramine (Benadryl), and/or steroids which may include solumedrol or prednisone. Tylenol is given by mouth, and Benadryl and steroids are given either by vein (over 10-15 minutes) or by mouth.

The combination of ATG and radiation will weaken your immune system. A weakened immune system may help to allow your body to "accept" donor cells, and it may decrease the chance of your body rejecting the cells.

If your diagnostic biopsy showed that a certain protein was found on your tumor cells, you may also receive rituximab therapy. If you are eligible for rituximab treatment, you will receive the drug once a week for 4 weeks. You will receive rituximab through the central venous catheter or through a vein over 6-8 hours. The first dose will be given on an outpatient basis at 13 days before the stem cell transplant. The next 3 doses may be given in the hospital or on an outpatient basis. You will receive rituximab 6 days before the transplant, and then 1 and 8 days after the transplant. Tylenol and steroids will be given before the rituximab to try to prevent an allergic reaction.

You will be given tacrolimus to try to prevent graft versus host disease (when the donor's immune cells react against the recipient's body, attacking the recipient's cells and tissues). You will receive tacrolimus either through the central venous catheter (over 24 hours each time) or by mouth starting 3 days before the stem cell transplant. You will continue receiving tacrolimus as long as your doctor feels it is necessary, which could be anywhere from about 3 months to several years. This will depend on factors such as whether or not you have graft versus host disease, how many donor cells are in your blood, and the status of your disease.

Cellcept (MMF) will also be given to try to prevent graft versus host disease, starting 1 day after the transplant and continuing through Days 28-42 after the transplant. The MMF will be given twice a day through the central venous catheter over 2 hours, or by mouth.

After the pre-transplant treatments and testing are finished, you will have the blood stem cell transplant. Blood stem cells from a donor will be infused over about 1 hour through your central venous catheter. This can be done while you are in the hospital or on an outpatient basis at M. D. Anderson. Steroids and Benadryl will be given through the catheter before the stem cell transplant to try to prevent an allergic reaction. The catheter will be removed once you no longer need to be given fluids, blood products, and other treatments through the catheter for graft versus host disease. This may take anywhere from 3 months after the transplant to several years.

You will have additional blood (about 2 tablespoons) drawn, bone marrow aspirations and biopsies, chest CT scans, and/or chest x-rays performed as needed to check the effects of the transplant. You will have transfusions of blood and platelets as needed, and you will have to sign a separate consent document for these transfusions.

Blood (about 1 tablespoon each time) will also be drawn at least 2-3 times a week for at least 100 days after the transplant, or longer if the study doctor feels it is necessary.

Treatment will be given in the hospital or an outpatient basis at M. D. Anderson. You may need to stay in the hospital for 3-4 weeks. You will be taken off the study if your disease gets worse.

This is an investigational study. The FDA has approved the drugs used in this study. Their use together in this study is investigational. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Age up to 70 years.
* Patients with lymphoid malignancies (primary refractory or recurrent) beyond first remission or unresponsive to therapy and not eligible for protocols of higher priority. Patients should have had at least a partial remission or have stable disease with prior chemotherapy. Patients with bulky disease (greatest dimension > 5 cm by radiographic or clinical examination are not eligible).
* Adequate renal function, as defined by serum creatinine <1.8 mg/dL.
* Adequate hepatic function, as defined by SGPT <3 times upper limit of normal; serum bilirubin and alkaline phosphatase <3 times upper limit of normal.
* Adequate pulmonary function with Forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and Carbon Monoxide Diffusing Capacity (DLCO) >35% of expected corrected for hemoglobin. Exceptions may be allowed for patients with pulmonary involvement after discussing with Principal Investigator.
* Adequate cardiac function with left ventricular ejection fraction >35%. No uncontrolled arrhythmias or symptomatic cardiac disease.
* Zubrod performance status <2
* Patients must have an human leukocyte antigens (HLA) matched, or one A, B, C, DR, or DQ mismatched related or unrelated donor (by high resolution typing). Donor must be willing to donate peripheral blood progenitor cells.
* Patient should be willing to participate in the study by providing written consent.
* Negative beta human chorionic gonadotrophin (hCG) test in a woman of child bearing potential (defined as not post menopausal for 12 months or no previous surgical sterilization).

Exclusion Criteria:

* Patients with active central nervous system (CNS) disease.
* Evidence of acute or chronic active hepatitis or cirrhosis.
* Uncontrolled infection, including Hepatitis B, C, Human immunodeficiency virus (HIV) or human T-cell lymphotropic virus type 1 (HTLV-1) infection.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chitra M. Hosing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 14, 2006 to October 15, 2008. All patients were registered at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Radiation + Chemotherapy + BSCT
Started | 20
Completed | 19
Not Completed | 1
Not completed — Progressive shortness of breath | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation + Chemotherapy + BSCT
Number analyzed (Participants) | 20
Age Continuous [Median (Full Range); unit: years] | 30 [20 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Composite Success Rate
Description: Defined as the proportions of the patients who are alive at day 100, are without Grade 3-4 Graft Graft-versus-host disease (GVHD), without Grade 4 toxicity (unrelated to infection) and have engrafted. Toxicity grades according to Common Toxicity Criteria (CTC) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0.
Time Frame: Baseline to Day 100, assessment at Day 100
Population: Analysis was per protocol. One participant was inevaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | Radiation + Chemotherapy + BSCT
Number analyzed (Participants) | 19
Percentage of participants
  Engraftment | 100
  Acute GvHD | 75
  alive at 100 days | 84

ADVERSE EVENTS:
Time Frame: 2 year, 5 months
Arm/Group | Radiation + Chemotherapy + BSCT
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation + Chemotherapy + BSCT (N=19)
increased bilrubin (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation + Chemotherapy + BSCT (N=19)
diarrhea (Gastrointestinal disorders) | 1 (1)
low blood pressure (Cardiac disorders) | 7 (7)
dysrhythmias (Cardiac disorders) | 1 (1)
tachycardia (Cardiac disorders) | 4 (4)
edema (Cardiac disorders) | 5 (5)
arterial (Cardiac disorders) | 2 (2)
other cardiac (Cardiac disorders) | 5 (5)
pain (Cardiac disorders) | 2 (2)
pericardial (Cardiac disorders) | 1 (1)
other endocrine (Endocrine disorders) | 3 (3)
fatigue (General disorders) | 7 (7)
rigors (General disorders) | 2 (2)
other general disorders (General disorders) | 7 (7)
fever (General disorders) | 7 (7)
nausea (Gastrointestinal disorders) | 9 (9)
Gastrointestinal other (Gastrointestinal disorders) | 13 (13)
diarrhea (Gastrointestinal disorders) | 5 (5)
Anorexia (Gastrointestinal disorders) | 1 (1)
increased creatinine (Renal and urinary disorders) | 5 (5)
bleeding (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)
cystitis (Renal and urinary disorders) | 3 (3)
pain (Gastrointestinal disorders) | 3 (3) — abdominal
increased Alkaline phosphatase (Hepatobiliary disorders) | 7 (7)
increased ALT (Hepatobiliary disorders) | 9 (9) — Alanine aminotransferase (ALT or SGPT)
increased biblrubin (Hepatobiliary disorders) | 5 (5)
increased LDH (Hepatobiliary disorders) | 3 (3)
infection (Infections and infestations) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
hypermagesium (Metabolism and nutrition disorders) | 4 (4)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
metabolic other (Metabolism and nutrition disorders) | 1 (1)
motor (Musculoskeletal and connective tissue disorders) | 3 (3)
headache (Nervous system disorders) | 9 (9)
other neruologic (Musculoskeletal and connective tissue disorders) | 6 (6)
insomnia (Nervous system disorders) | 2 (2)
neurologic mood (Nervous system disorders) | 4 (4)
eye pain (Eye disorders) | 2 (2)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 5 (5)
rash (Skin and subcutaneous tissue disorders) | 7 (7)
skin other (Skin and subcutaneous tissue disorders) | 3 (3)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to financial support.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No